CLINICAL TRIAL: NCT06497075
Title: The Feasibility and Acceptability of the Co-administration of Ivermectin and Albendazole vs Albendazole Alone, in the Frame of Mass Drug Administration to School-aged Children in Uganda: A Small-scale Implementation Pilot Study
Brief Title: Co-administration of IVM and ALB in School-based Deworming in Uganda
Acronym: FACE-ITpilot
Status: Completed | Type: Observational
Sponsor: Jennifer Keiser (Other)
Collaborators: Vector Borne & Neglected Tropical Disease Control Division, Ministry of Health, Uganda (Unknown); Makerere University (Other)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Prof. Dr., Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Other Study IDs: 2283p
Record Dates: First submitted 2024-06-26; First posted 2024-07-11 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Helminthiasis; Intestinal Worms
Keywords: soil-transmitted helminths; ivermectin; deworming; albendazole
MeSH Terms: conditions — Helminthiasis | interventions — Albendazole; Ivermectin

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Albendazole only: Schoolchildren aged 5-14 years of 10 schools randomized to receive the standard deworming treatment of a single dose of albendazole 400mg.
  Interventions: Drug: Albendazole 400mg
- Ivermectin and albendazole: Schoolchildren aged 5-14 years of 10 schools randomized to receive the combination treatment of a single dose of ivermectin 200ug/kg (according to height category using a dose-pole) plus albendazole 400mg.
  Interventions: Drug: Albendazole 400mg; Drug: Ivermectin 3 MG

INTERVENTIONS:
Drug: Albendazole 400mg — Single oral dose of Albendazole 400mg tablet
  Other Names: Zentel
Drug: Ivermectin 3 MG — Generic ivermectin 3mg tablets given as a single oral dose of 200ug/kg using a dose-pole (height categories: 90-119 cm: 1 tablet , 120-140 cm: 2 tablets, 141-158 cm: 3 tablets or > 158 cm: 4 tablets)
  Other Names: Mectizan; Stromectol
  Groups: Ivermectin and albendazole

SUMMARY:
The goal of this small-scale implementation research pilot study is to assess the feasibility and acceptability of the co-administration of ivermectin (IVM) and albendazole (ALB) compared to albendazole alone during school-based mass drug administration in Uganda. The study will target up to 10,000 school-aged children from 20 schools in Kabale and Kisoro districts in South-Western Uganda.

The main questions it aims to answer are:

* How feasible is the introduction of co-administered IVM plus ALB in the routine school-based deworming campaign in terms of training, material and processes?
* How well do beneficiary communities (pupils, parents) and implementers (teachers, health workers) accept the new treatment scheme and what are potential barriers and enablers for uptake?
* What are common implementation-related costs that can inform the methodology to estimate monetary and non-monetary costs as well as performance of the two treatment arms for the future cost-effectiveness analysis?

The study employs a cross-sectional mixed-method design (we will collect qualitative and quantitative data) to evaluate the feasibility and acceptability of co-administering IVM and ALB versus ALB alone in routine school-based mass drug administration. Assessments will take place during and after the drug distribution to document the implementation process and evaluate experiences made by the different stakeholders (e.g. children, parents, teachers, health workers):

* The implementation activities start with a training of all implementers at district level who will also undergo a pre- and post-training knowledge assessment.
* Schoolchildren aged 5-14 years will receive a single dose of ALB alone or co-administered ALb (400mg) and IVM (200µg/kg; as determined by height category on a dose pole) by health workers at school. 1-2 weeks post-distribution a subsample of 19 children per school will be invited to answer to questionnaires administered by social science researchers.
* Implementers will administer the treatments and document all distribution-related aspects during the campaign under supervision of the routine staff. Researchers will conduct additional monitoring and evaluation in order to assure data quality and provide support in performance assessment and cost evaluation.
* Beneficiaries (parents) and implementers will be asked to take part in focus group discussions and questionnaire interviews one week after the drug distribution.

ELIGIBILITY:
* School-aged children (5-14 years) of the selected schools
* Written informed consent from the participant's parents/caretakers and assent (for children aged 8 years and older) from the participant him/herself or written informed consent from the school teacher (for children attending schools receiving routine albendazole deworming)
* No signs of major acute or chronic illness
* No known allergy to study medication (i.e. benzimidazoles or ivermectin)

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Study population receiving intervention: All eligible school-aged children (5-14 years) from 20 pre-selected schools present in the school at the day of the treatment campaign, will be treated with the respective single or combination treatment regimen depending on the treatment arm under which the schools fall.
  * Study population of post-distribution social science study: Subsamples of treated schoolchildren, parents of school-aged children of the respective study schools, teachers involved in distribution, health workers involved in distribution.
Sampling Method: Non-Probability Sample
Enrollment: 8767 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-10-19 (Actual)

PRIMARY OUTCOMES:
Feasibility of IVM + ALB introduction | Documentation before, during and up to 12 weeks after the drug distribution
  Feasibility will be assessed using quantitative and qualitative data sources for the following performance and process indicators:
  * Reported therapeutic coverage (proportion)
  * Programme reach (proportion)
  * Compliance rate (children that ingested drugs divided by the total number of children who got offered the drugs)
  * Reasons for not offering the drugs (non-eligibility)
  * Reasons for not swallowing the drugs (refusal)
  * Reported safety: Number, type and severity of adverse events recorded
  * Incremental time needs for IVM-ALB co-administration
  * Additional training needs
  * Incremental staff needs
  * Drug logistics (tablet balance)
  Short and structured training evaluation questionnaires will be administered to teachers and health workers directly after training and cover aspects on (i) drug dosing including dose-pole utilization, (ii) identification of non-eligible populations, (iii) documentation processes and (iv) drug information (including safety)

SECONDARY OUTCOMES:
Acceptability and barriers & enablers to introduction of IVM-ALB co-administration (recipient perspective) | 1-2 weeks after drug distribution
  Qualitative data on acceptability of the intervention from a recipient perspective (parents) will be collected trough FGDs that will cover:
  * Current knowledge about STHs: transmission, health impact, prevention and treatment
  * Prior knowledge of MDA activities and related experiences
  * Potential enabling factors for willingness of parents to let their children participate in MDA
  * Potential barriers for acceptance of parents for their child's participation in MDA
  Quantitative data on acceptability of the intervention from a recipient perspective (schoolchildren) will be collected through structured interviews using Likert scale questions (5-point scale from strongly disagree to strongly agree) and cover aspects on:
  * Attitudes towards treatment
  * Convenience of taking the treatment
  * Self-reported willingness and understanding for need of treatment
  * Self-reported satisfaction with the treatment and procedures of the campaign
Potential incremental costs related to IVM-ALB co-administration | Documentation before, during and up to 12 weeks after the drug distribution
  The following cost components related to the activities required to implement the interventions will be included in the analysis:
  * Medicine Procurement and Distribution: Costs associated with purchasing and distributing albendazole and ivermectin.
  * Stationary and Supplies: Costs related to necessary materials for documentation and record-keeping.
  * Transport: Costs involved in transporting medicines and supplies to the designated MDA locations.
  * Allowances: Allowances provided to personnel involved in the implementation.
  * Training Costs: Expenses associated with training personnel on the co-administration protocol.
  * Personnel Time: Costs of personnel time dedicated to delivering interventions.
Acceptability and barriers & enablers to introduction of IVM-ALB co-administration (provider perspective) | 1-2 weeks after drug distribution
  Qualitative data on acceptability of the intervention from a provider perspective (teachers and health workers) will be collected trough FGDs and KIIs and will cover:
  * Current knowledge about STHs: transmission, health impact, prevention and treatment
  * Prior involvement in any MDA activities and related experiences
  * Post-distribution training evaluation
  * Potential enabling factors for willingness and barriers for acceptance of parents to let their children participate in MDA
  Quantitative data on acceptability of the intervention from a provider perspective will be collected through structured interviews using Likert scale questions (5-point scale from strongly disagree to strongly agree) and cover:
  * Attitudes towards treatment
  * Convenience of distributing the treatment and satisfaction with training
  * Observed willingness and understanding for need of treatment
  * Observed satisfaction with the treatment and procedures of the campaign

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Keiser, Prof., Principal Investigator — Swiss Tropical & Public Health Institute
Locations (2):
- Uganda (2):
  - Makerere University, College of Humanities and Social Sciences, Kampala
  - Vector Borne & Neglected Tropical Disease Control Division, Ministry of Health, Kampala

IPD SHARING:
Plan to Share IPD: No
There is a data sharing agreement between Swiss TPH, Uganda MoH and Makerere University in place. Data may be shared with other researchers upon request.